CLINICAL TRIAL: NCT02221947
Title: A Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Preliminary Safety, Efficacy, Pharmacokinetics and Pharmacodynamics of Bryostatin 1 in Patients With Alzheimer's Disease
Brief Title: Study to Evaluate the Preliminary Safety, Efficacy, PK and PD of Bryostatin 1 in Patients With Alzheimer's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Part 2 of study replaced by NTRP-101-202, assessing 3 doses of bryostatin.
Sponsor: Neurotrope Bioscience, Inc. (Industry)
Collaborators: Blanchette Rockefeller Neurosciences Insitute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTRP101-201
Record Dates: First submitted 2014-07-02; First posted 2014-08-21 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; bryostatin; PKC epsilon
MeSH Terms: conditions — Alzheimer Disease | interventions — bryostatin 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bryostatin 1 (Active Comparator): single dose of 25 μg/m2 bryostatin, intravenous infusion over 1 hour
  Interventions: Drug: Bryostatin 1
- placebo (Placebo Comparator): single dose of placebo, intravenous infusion over 1 hour
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bryostatin 1 — 25 μg/m2 bryostatin 1, single dose via intravenous infusion over 1 hour.
  Arms: Bryostatin 1
Drug: Placebo — Placebo, single dose via intravenous infusion over 1 hour.
  Arms: placebo

SUMMARY:
This study is being done to evaluate the safety, tolerability and potential effectiveness of a new investigational drug, bryostatin 1, in patients with Alzheimer's disease (AD).

DETAILED DESCRIPTION:
This study is a single center, randomized, double-blind, placebo-controlled, parallel groups trial in patients with AD. Each subject enrolled in the trial will be randomized to receive a single IV dose of 0 (placebo) or 25 μg/m2 bryostatin. A total of 15 subjects (5 in the placebo arm and 10 in the treatment arm) will be enrolled in the study. The study consists of screening evaluations and on study evaluations divided into two segments, an inpatient segment and an outpatient segment. The four-day inpatient segment will consist of baseline evaluations and a 1-hour IV infusion of study drug followed by evaluations at multiple evaluations over the first 72 hrs post dose. During the outpatient segment, patients will be followed for AEs and have a final evaluation at 2 weeks post dose and a 4-week telephone safety follow up. Evaluations will include safety, efficacy, pharmacokinetics, and pharmacodynamics as assessed by PKC activity

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 50 - 85 yrs. Females are non-childbearing potential
* Patient must have a cognitive deficit present for at least 1 year and meet diagnostic criteria for probable Alzheimer's Disease Dementia by NIA-AA criteria or prodromal Alzheimer's Disease
* Mini Mental State Exam score of 16-26
* Ability to walk, at least with an assistive device
* Vision and hearing sufficient to comply with testing
* Normal cognitive and social functioning prior to onset of dementia, with evidence of progressive symptoms from patient or informant
* Consistent caregiver to accompany patient to visits
* Sufficient basic education to be able to complete the cognitive assessments
* Living outside an institution

Exclusion Criteria:

* Dementia due to any condition other than AD, including vascular dementia
* Significant neuroimaging abnormalities, previously known or discovered on screening MRI scan,
* Evidence of clinically significant unstable cardiovascular, renal, hepatic, gastrointestinal, neurological, or metabolic disease within the past 6 months
* Use of any drug within 14 days prior to randomization unless the dose of the drug and the condition being treated have been stable for at least 30 days and are expected to remain stable during the study
* Use of tobacco products or nicotine-containing products within 3 months before Day 1
* Use of high dose vitamin E, or valproic acid
* Any medical or psychiatric condition that may require medication or surgical treatment during the study
* Life expectancy less than 6 months
* Use of an investigational drug within 2 months prior to the screening visit
* Clinically significant neurological disease other than AD
* Major depression, alcohol or drug dependence or suicidality
* Psychotic episodes requiring hospitalization or antipsychotic therapy for more than 2 weeks within the past 10 years, not linked to AD
* Agitation sufficient to preclude participation in this trial
* Epilepsy or anti-epileptic drug therapy
* Abnormal laboratory tests that might point to another etiology for dementia;
* Acute or poorly controlled medical illness
* Likelihood, according to clinical judgment, of being transferred to a nursing home within 6 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hakop Gevorkyan, MD, MBA, Principal Investigator — California Clinical Trials Medical Group
Locations (1):
- California Clinical Trials Medical Center, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bryostatin 1 | Placebo
Started | 6 | 3
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bryostatin 1 | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (8.04) | 70.7 (7.23) | 71.9 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Evaluate the safety and tolerability of bryostatin 1 (hereinafter referred to as bryostatin) in patients with Alzheimer's Disease (AD) following a single intravenous (IV) dose.
Time Frame: Within 2 weeks of study drug dosing
Measure: Number; unit: event
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 6 | 3
event
  Dizziness | 0 | 1
  Headache | 1 | 1
  Rash Papular | 0 | 1

2. Primary Outcome: Preliminary Efficacy of a Single Dose of Bryostatin in the Treatment of Patients With AD
Description: Hopkins Verbal Learning Test - Revised (HVLT-R) delayed recall; change from baseline. HVLT consists of a 12-item word list drawn from 3 semantic categories, presented in 3 learning trials. Score range = 0-12. The lower the number, the more impaired.
  Repeatable Battery of Assessments for Neuropsychological Status (RBANS) figure recall; change from baseline. Total Score Range: 0-20. Each portion of the drawing is scored 1 point for correctness and completeness and 1 point for being placed properly in relation to the rest of the drawing. Drawing and placement scores are summed for the item total. To obtain subtest total score, the drawing and placement scores are summed for each item. The lower the number, the more impaired.
Time Frame: 48 hours post start of study drug infusion
Measure: Mean (Standard Deviation); unit: units on a scale, change from baseline
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 6 | 3
units on a scale, change from baseline
  HVLT-R at 48hrs (change from baseline) | 1.3 (2.16) | 3.7 (1.15)
  RBANS figure recall at 48hrs (CBL) | 4.5 (4.14) | 6.7 (3.06)

3. Secondary Outcome: Preliminary Efficacy of a Single Dose of Bryostatin in the Treatment of Patients With AD
Description: HVLT-R (Hopkins Verbal Learning Test-Revised™) delayed recall (change from baseline). A 12-item word list: 3 learning trials. Score range = 0-12. The lower the number, the more impaired.
  Repeatable Battery of Assessments for Neuropsychological Status (RBANS) figure recall; change from baseline. Score Range: 0-20. The lower the number, the more impaired. Digit Symbol Coding (observed), Score range: 0-125. The lower the number, the more impaired.
  Clinical Dementia Rating- Sum of Boxes (CDR-SB, observed). Sum of 6 investigated domains (Memory, Orientation, Judgment and Problem Solving, Community Affairs, Home and Hobbies, Personal Care). Each subtest range is 0-3; Sum of all 6 subtest scores gives total CDR-SB score (range= 0-18).The higher the number, the more impaired.
  Mini Mental State Exam, version 2 (MMSE-2), change from baseline. The MMSE-2 measures aspects of cognitionon a scale of 0-30. Lower scores indicate greater cognitive impairment.
Time Frame: Specified timepoints within 2 weeks post study drug infusion
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo: single dose via intravenous infusion over 1 hour.
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 6 | 3
units on a scale
  HVLT-R 24hr Delayed Recall (change from baseline) | 0.5 (3.27) | 1.3 (2.52)
  HVLT-R 2 Wks Delayed Recall (change from baseline) | 0.3 (1.63) | 2.3 (2.52)
  RBANS 24hr Figure Recall (change from baseline) | 4.7 (4.76) | 6.0 (2.65)
  RBANS 2 Wks Figure Recall (CBL) | 4.2 (5.60) | 7.3 (3.06)
  HVLT-R delayed recall of stimuli at 48hr (CBL) | -1.2 (1.17) | 2.7 (2.08)
  Digit Symbol Coding baseline (observed) | 32.2 (9.13) | 42.3 (12.50)
  Digit Symbol Coding 24hrs post start of infusion | 36.0 (10.75) | 49.0 (4.58)
  Digit Symbol Coding 48hrs post start of infusion | 37.3 (11.64) | 53.7 (4.73)
  Digit Symbol Coding 2 wks post start of infusion | 38.3 (7.61) | 52.7 (6.66)
  CDR, CDR-SB baseline (observed) | 1.3 (0.98) | 0.7 (0.29)
  CDR, CDR-SB 2wks (observed) | 1.5 (1.00) | 0.7 (0.29)
  MMSE-2 3hrs post start of inf (change) | 1.8 (1.72) | -1.0 (2.65)
  Digit Symbol Coding baseline (observed) | 32.2 (9.13) | 42.3 (12.50)
  Digit Symbol Coding 3hrs post start of inf (observ | 32.7 (6.86) | 45.3 (11.50)
  MMSE-2 at 72hrs (change from Baseline) | 2.6 (1.52) | 3.3 (2.52)
  MMSE-2 at 2wks (change from Baseline) | 3.3 (1.86) | 4.7 (1.15)

4. Other Pre Specified Outcome: Pharmacokinetic Parameters of Bryostatin.
Description: Preliminary evaluation of pharmacokinetics and pharmacodynamics (Cmax, Tmax, AUClast).
Time Frame: Bryostatin plasma concentration pre-dose and at 15 min, 30 min, 1 hr, 1.5 hr, 2hr, 3hr and 6rs post dose.
Population: Subjects who received a single dose of 25 μg/m2 bryostatin, intravenous infusion over 1 hour (PK population)
Measure: Mean (Standard Deviation); unit: bryostatin plasma concentration (ng/mL)
Arm/Group | Bryostatin 1 | Placebo
Number analyzed (Participants) | 6 | 0
bryostatin plasma concentration (ng/mL)
  predose Bryostatin Plasma Concentration (ng/mL) | 0.0 (0.0) |
  Concentration 15 min post (ng/mL) | 0.880 (0.133) |
  Concentration 30 min post (ng/mL) | 0.941 (0.168) |
  Concentration 1 hr post (ng/mL) | 1.04 (0.309) |
  Concentration 1.5 hrs post (ng/mL) | 0.181 (0.148) |
  Concentration 2 hrs post (ng/mL) | 0.0702 (0.109) |
  Concentration 3 hrs post (ng/mL) | 0.0 (0.0) |
  Concentration 6 hrs post (ng/mL) | 0.0 (0.0) |
  Cmax (ng/mL) | 1.09 (0.246) |
Statistical Analysis 1: Comparison: Bryostatin 1; Bryostatin plasma concentration: mean Tmax (h); Test type: Other; mean Tmax(h) = 0.920 — SD=0.206
Statistical Analysis 2: Comparison: Bryostatin 1; Bryostatin plasma concentration AUC0-last (h*ng/mL); Test type: Other; mean (h*ng/mL) = 1.05 — SD=0.330

ADVERSE EVENTS:
Time Frame: Adverse event collection began 28 days prior to dosing and continued until 4 weeks after dosing. Ongoing AEs were followed until resolved or stabilized.
Arm/Group | Bryostatin 1 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 1/6 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bryostatin 1 (N=6) | Placebo (N=3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot disclose trial results without permission from sponsor.